CLINICAL TRIAL: NCT04469699
Title: Controlled Clinical Trial to Evaluate the Safety and Efficacy of Stereotactical Photodynamic Therapy With 5-aminolevulinic Acid (Gliolan®) in Recurrent Glioblastoma
Brief Title: Stereotactical Photodynamic Therapy With 5-aminolevulinic Acid (Gliolan®) in Recurrent Glioblastoma
Acronym: NOA11
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other); photonamic GmbH & Co. KG (Industry); medac GmbH (Industry); LifePhotonic GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKM12_0017; 2015-002727-25 (EudraCT Number)
Record Dates: First submitted 2020-05-12; First posted 2020-07-14 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Glioblastoma Multiforme, Adult
MeSH Terms: conditions — Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): Stereotactic biopsy followed by stereotactical photodynamic therapy
  Interventions: Drug: Stereotactic biopsy followed by stereotactical photodynamic therapy with 5-aminolevulinic acid
- Control arm (Other): Stereotactic biopsy
  Interventions: Procedure: Stereotactic biopsy

INTERVENTIONS:
Drug: Stereotactic biopsy followed by stereotactical photodynamic therapy with 5-aminolevulinic acid — 5-ALA HCl orally (20 mg/kg bw) 3,5-4,5 hours prior to induction of anaesthesia for stereotactic biopsy followed by stereotactical photodynamic therapy. All patients will receive further treatment of recurrent glioblastoma at the investigator´s discretion (best possible care).
  Other Names: Gliolan, 5-aminolevulinic acid
  Arms: Treatment arm
Procedure: Stereotactic biopsy — Stereotactic biopsy. All patients will receive further treatment of recurrent glioblastoma at the investigator´s discretion (best possible care).
  Arms: Control arm

SUMMARY:
In this multicenter, randomized, non-blinded trial the efficacy and safety of stereotactical photodynamic therapy with 5-aminolevulinic acid will be investigated in 106 patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Age 18 - 75 years
3. Karnofsky Performance Score (KPS) of ≥60 %
4. Radiologically suspected diagnosis (according to RANO criteria) of the first recurrence of a glioblastoma located in the cerebral hemisphere including insular and diencephalon. Tumors in the brain stem are excluded. First MRI with signs of first recurrence (radiologic RANO criteria for disease progression) within 8 weeks prior to Informed Consent. Not necessarily identical to primary tumor location
5. Single or single progressive contrast-enhancing lesion on MRI, largest diameter not more than 2.5 cm
6. For female and male patients of reproductive potential: Willingness to apply highly effective contraception (Pearl index <1) during the entire study

Exclusion Criteria:

1. Multifocal disease > 2 locations
2. Patients with significant non-enhancing tumor portions
3. Previous treatment of recurrence
4. Other malignant disease except basalioma
5. Hypersensitivity against porphyrins or Gliolan® or Fluorethylenpropylen (FEP )
6. Porphyria
7. HIV infection, active Hepatitis B or C infection
8. Bone marrow reserve:

   * white blood cell (WBC) count <2000/μl,
   * platelets <100000/μl,
9. Liver function:

   * total bilirubin > 1.5 times above upper limit of normal range (ULN)
   * alanine transaminase (ALT) and aspartate transaminase (AST) > 3 times ULN
10. Renal function:

    - creatinine > 1.5 times ULN
11. Blood clotting:

    - Quick/INR or PTT out of acceptable limits
12. Conditions precluding MRI (e.g. pacemaker)
13. Past medical history of diseases with poor prognosis, e.g. severe coronary heart disease, heart failure (NYHA III/IV), severe poorly controlled diabetes, immune deficiency, residual deficits after stroke, severe mental retardation or other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
14. Any active infection (at the discretion of the investigator)
15. Any psychological, cognitive, familial, sociological or geographical condition that, in the investigator's opinion, compromises the patient's ability to understand the patient information, to give informed consent or to comply with the trial protocol
16. Previous antiangiogenic treatment
17. Participation in another interventional clinical trial during this trial or within 4 weeks before entry into this trial.
18. Pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | through study completion (at least 1.5 years and a maximum of 5 years) or until progression or death
  Progression free survival (PFS) measured as time from the day of randomization until diagnosis of progressive disease as determined by MRI according to RANO criteria (Response Assessment in Neuro-Oncology Criteria) or death from any cause

SECONDARY OUTCOMES:
6-month PFS rate | for each patient up to 6 months after randomization or until progression has occurred
  Progression free survival (PFS) measured as time from the day of randomization until diagnosis of progressive disease as determined by MRI according to RANO criteria or death from any cause
Overall survival (OS) | through study completion (at least 1.5 years and a maximum of 5 years) or until death
  Overall survival (OS) measured as time from the day of randomization until death
Progression free time | through study completion (at least 1.5 years and a maximum of 5 years) or until progression
  Progression free time as time from the day of randomization until progressive disease (death is regarded as censored)
12-month OS rate | for each patient up to 12 months after randomization or until death
  Overall survival (OS) measured as time from the day of randomization until death
Absolute changes from baseline in contrast medium volume uptake from the MRI performed 48 hours after randomization on, and during any MRI performed thereafter to monitor for disease progression | Baseline, 26 - 48 hours after stereotactic procedure, 1 month after randomization and then every 2 months, 1.5 years after randomization or at disease progression, and then every 3 months until end of entire study (up to 5 years) or progression
48h response rate on MRI (Complete Remission, Partial Remission, Stable Disease) after treatment with iPDT (interstitial photodynamic therapy) | 26 - 48 hours after stereotactic procedure in patients treated with interstitial photodynamic therapy (iPDT)
  Response is assessed according to the RANO criteria
If a PET (positron emission tomography) was performed less than 2 weeks apart from an MRI: Consistency of both procedures with regard to the region of interest (ROI) | Baseline, 26 - 48 hours after stereotactic procedure, 1 month after randomization and then every 2 months, 1.5 years after randomization or at disease progression and then every 3 months until end of entire study (up to 5 years) or progression
Change in KPS (Karnofsky Performance Score) | Baseline, 26 -48 hours after stereotactic procedure, upon discharge or 7 days after stereotactic procedure, 1 month after randomization and then every 2 months until 1.5 years after randomization or disease progression
  Minimum value: 0, maximum value: 100. A higher value means a better outcome.
Change in NIHSS (National Institutes of Health Stroke Scale) | Baseline, 26 -48 hours after stereotactic procedure, upon discharge or 7 days after stereotactic procedure, 1 month after randomization and then every 2 months until 1.5 years after randomization or disease progression
  Minimum value: 0, maximum value: 42. A higher value means a worse outcome.
Change in MMSE (Mini-Mental State Examination) | Baseline, 26 -48 hours after stereotactic procedure, upon discharge or 7 days after stereotactic procedure, 1 month after randomization and then every 2 months until 1.5 years after randomization or disease progression
  Minimum value: 0, maximum value: 30. A higher value means a better outcome.
Brain edema as assessed by MRI within 26 to 48 h after stereotactic surgery | 26 to 48 hours after stereotactic intervention
Frequency of Adverse Events | over the entire study period of each patient (at least 1.5 years and a maximum of 5 years)
Change in the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Core Quality of Life Questionnaire) score during study participation | Baseline, at discharge or 7 days after intervention, 1 month after randomization and then every 2 months, 1.5 years after randomization or at disease progression and then every 3 months until end of entire study (up to 5 years) or progression
Change in the EORTC QLQ-BN20 module (European Organisation for Research and Treatment of Cancer Quality of Life Brain Cancer Module) score during study participation | Baseline, at discharge or 7 days after intervention, 1 month after randomization and then every 2 months, 1.5 years after randomization or at disease progression and then every 3 months until end of entire study (up to 5 years) or progression

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stummer, Univ.-Prof. Dr. med., Principal Investigator — University Hospital Muenster, Klinik und Poliklinik für Neurochirurgie
Locations (4):
- Germany (4):
  - Medizinische Fakultät Carl Gustav Carus, Klinik und Poliklinik für Neurochirurgie, Dresden
  - Universitätsklinikum Düsseldorf, Klinik für Neurochirurgie, Abteilung Funktionelle NC & Stereotaxie, Düsseldorf
  - Universitätsklinikum Essen, Klinik für Neurochirurgie und Wirbelsäulenchirurgie, Essen
  - Universitätsklinikum Münster, Klinik und Poliklinik für Neurochirurgie, Münster

IPD SHARING:
Plan to Share IPD: No